CLINICAL TRIAL: NCT00516594
Title: The Effect of Altering Colonic Microflora After Fiber (FOS) Consumption on Blood Lipids Risk Factors for Heart Disease in Healthy "Normal" and Hyperlipidemic Subjects
Brief Title: The Effect of Altering Colonic Microflora After Fiber (FOS) Consumption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); Orafti Group (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB 205UC
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Hyperlipidemia; Cardiovascular Disease; Diet Therapy
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases | interventions — Diet; Soybean Proteins

INTERVENTIONS:
Procedure: Diet with polyfructans and viscous fibers or soy protein

SUMMARY:
Our antibiotic studies indicated that cholesterol lowering was seen when fecal bifidobacterial counts were increased. Due to the dangers associated with prolonged antibiotic use we have been funded by the Heart and Stroke Foundation to see if gut bacteria can be modified by non-antibiotic means. Inulin a dietary fiber found in artichokes, chicory, leaks, onion, etc., (which also produces flatulence) has been shown to increase bifidobacteria and also appears to lower serum cholesterol. We will therefore test the fiber to determine its effectiveness in lowering serum cholesterol and whether it can be used to maximize the cholesterol-lowering effects of soy protein foods and viscous fiber foods (e.g. oats and psyllium).

DETAILED DESCRIPTION:
Design: Studies will be three phase randomized crossover design with all subjects undergoing all three phases. Each phase will be one month in duration with at least 2-4 weeks washout between phases.

General Protocol: Both dietary studies (Study 1 fiber plus polyfructans; and Study 2 soy plus polyfructans) will follow the same general protocol. Supplements and measurements will differ between studies. Diets will be self-selected low-fat diets throughout (<7% of total energy as saturated fat and, <200 mg/d dietary cholesterol). Supplements will be provided at weekly intervals. At the start and at two weekly intervals during the study body weight, blood pressure and fasting bloods will be taken together with 24h urine and 4-day fecal collections and samples for fecal microbiology to be obtained during week 4. Treatments: Both studies will involve a control diet which will be an NCEP step 2 diet (low in saturated fat and dietary cholesterol) with 10-20 g inulin. Study 1 subjects will take 10-15 g viscous fiber foods with or without the fructan. Study 2 subjects will take 30-40 g soy protein foods with or without the fructan (please see Table 1). The supplements will be provided as foods: oat bran bread to be taken with meals and as snacks during Study 1 and soy protein to be taken in soy beverage, soy hot dogs, burgers, tofu, etc., during Study 2.

Study Details: Subjects will come after a 12h overnight fast to the Risk Factor Modification Centre at St. Michael's Hospital immediately prior to commencement of each treatment phase and at weekly intervals during the course of each study period. Prior to the start of the study, subjects will be instructed on details of the study diet protocol. They will also be asked to maintain a constant level of physical activity throughout the course of the study. At all visits, body weight (in kg) will be obtained in indoor clothing, without shoes, and blood pressure will be taken twice in the dominant arm after subjects have been seated for at least 20 minutes. Height (in cm) will be recorded at the first visit. Throughout the study period, subjects will maintain their usual diet, which should be an NCEP step 2 diet (low saturated fat). Subjects will provide a fasting blood sample at week 0 and at weekly periods throughout the study. At weeks 0, and 4 seven-day food records will be collected. Subjects will also be weighed and seated blood pressure will be taken. Breath samples, 24h urine and 4-day fecal collections will be made at the beginning of the study and at the end of each study phase.

Diets: Initial dietary records prior to the start of the study together with instruction from the dietitian will ensure all subjects are on low fat (<7% of energy from saturated fat), low cholesterol diets (<200 mg/d), which they will maintain throughout the study. During the study subjects will collect their supplements at weekly intervals and return uneaten supplements. Subjects will be provided with self-tarring scales and diet history forms on which to record all food eaten together with the weights of all food items consumed during each study phase. These will be checked by the dietitian at weekly intervals to ensure compliance with the diet plan and to ensure there are no changes in body weight. Photocopies of the first week's diet record will be provided to each subject at the start of each phase to act as a dietary template and ensure consistency between studies. Compliance: This will be assessed by the return of uneaten supplements which will be weighed at the end of each phase and from the completed weekly check lists of supplements eaten and seven day diet records.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C > 4.1 mmol/L at recruitment
* living within a 40 km radius of St. Michael's Hospital

Exclusion Criteria:

* lipid lowering medications
* clinical or biochemical evidence of diabetes, renal or hepatic disease
* body mass index (BMI) >32 kg/m2
* antibiotic use within the last three months
* hormone replacement therapy
* smoking or significant alcohol intake (>1 drink/d)
* triglyceride level >4.0 mmol/L

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Total and LDL cholesterol, Total:HDl cholesterol ratio

SECONDARY OUTCOMES:
antropometrics: body weight, blood pressure, blood: triglycerides, fecal: SCFA and microbiology, breath: gases, urine: soy isoflavones, creatinine, urea, electrolytes

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PHD, DSc, Principal Investigator — University of Toronto and St. Michael's Hospital
Locations (1):
- Clinical Nutrition & Risk Factor Modification Centre, St. Michael's Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wong JM, Kendall CW, Marchie A, Liu Z, Vidgen E, Holmes C, Jackson CJ, Josse RG, Pencharz PB, Rao AV, Vuksan V, Singer W, Jenkins DJ. Equol status and blood lipid profile in hyperlipidemia after consumption of diets containing soy foods. Am J Clin Nutr. 2012 Mar;95(3):564-71. doi: 10.3945/ajcn.111.017418. Epub 2012 Feb 1. PMID 22301925